CLINICAL TRIAL: NCT01634243
Title: A Open-label Dose-ranging Study for SPM 962 in Parkinson's Disease Patients
Brief Title: A Dose-ranging Study for SPM 962 in Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-03-001
Record Dates: First submitted 2012-06-27; First posted 2012-07-06 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
Keywords: SPM 962; rotigotine; Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPM 962 (Experimental): SPM 962 transdermal patch
  Interventions: Drug: SPM 962

INTERVENTIONS:
Drug: SPM 962 — SPM 962 transdermal patch once a daily up to 36.0 mg/day
  Other Names: rotigotine

SUMMARY:
The primary objective of this trial is to establish the maximum maintenance dose of SPM 962 in patients with Parkinson's disease in a multi-center, uncontrolled, open-label study by conducting safety evaluation of each patient following once-daily transdermal doses of SPM 962 within a range of 4.5 to 36.0 mg. (The administration period will consist of a standard 8-week dose-titration period, 4-week dose-maintenance period, and a dose de-escalation period) Exploratory evaluation of each patient's maintenance dose will also be conducted with attention to patient safety. The relationship of pharmacokinetics, safety, and efficacy will also be examined.

ELIGIBILITY:
Inclusion Criteria:

* For subject with early and advanced Parkinson's disease

  * Subject diagnosed as having Parkinson's disease in accordance with "Diagnostic Criteria established by the Research Committee of MHLW-specified Intractable Neurodegenerative Diseases (1995)".
  * Subject is 30 and more and less than 80 years of age at the time of informed consent.
  * Gender and inpatient-outpatient status are not specified.
* For subject with early Parkinson's disease

  * Hoehn & Yahr stage 3 or less.
  * Subject who has not taken L-dopa within 28 days prior to initial administration of SPM 962.
* For subject with dvanced Parkinson's disease

  * Hoehn & Yahr stage 2-4.
  * Subject is on a stable dose of L-dopa with no change in daily dose or dosing regimen for at least 7 days prior to the initial treatment of SPM 962.
  * Subject has any of the following problematic symptoms; 1) Wearing off phenomenon 2) On and off phenomenon 3) Not well controlled with L-dopa due to adverse effect 4) Weakening of L-dopa efficacy.

Exclusion Criteria:

* Subject is on other dopamine agonist treatment within 7 days prior to the initial treatment. Subject is on cabergoline treatment within 14 days prior to the initial treatment.
* Subject has psychiatric symptoms, e.g. confusion, hallucination, delusion, excitation, delirium, abnormal behavior.
* Subject has orthostatic hypotension.
* Subject has a history of epilepsy, convulsion and other.
* Subject has a complication of serious cardiac disorder or has the history.
* Subject has arrhythmia and treated with class 1a antiarrhythmic drugs (e.g. quinidine, procainamide etc.) or class 3 antiarrhythmic drugs (e.g. amiodarone, sotalol etc.).
* At screening and baseline, subject develops serious ECG abnormality. Subjects has QTc-interval >450 msec at screening. Subject has QTc-interval >450 msec in males and >470 msec in females at baseline.
* Subject has congenital long QT syndrome.
* Subject has hypokalaemia.
* Subject has a total bilirubin >= 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or >= 100 IU/L).
* Subject has BUN >= 25 mg/dL or serum creatinine >= 2.0 mg/dl.
* Subject has a history of allergic reaction to topical agents such as transdermal patch.
* Subject is pregnant or nursing or woman who plans pregnancy during the trial.
* Subject is receiving therapy with prohibited drug specified in the study protocol.
* Subject has a history of pallidotomy, thalamotomy, deep brain stimulation or fetal tissue transplant.
* Subject has dementia.
* Subject is unable to give consent.
* Subject is participating in another trial of an investigational drug or done so within 6 months prior to the initial treatment.
* Investigator judges that subject is inappropriate as a study subject with other reasons.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2005-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (5):
- Japan (5):
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- Early-stage Parkinson's Disease: Subjects with early Parkinson's disease received SPM 962 transdermal patch
- Advanced Parkinson's Disease: Subjects with advanced Parkinson's disease received SPM 962 transdermal patch
Period: Overall Study
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Started | 21 | 43
Completed | 15 | 38
Not Completed | 6 | 5
Not completed — Adverse Event | 5 | 5
Not completed — Lack of Efficacy | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease | Total
Number analyzed (Participants) | 21 | 43 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (6.9) | 64.7 (7.6) | 64.6 (7.3)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 20 | 32
  >=65 years | 9 | 23 | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 29 | 41
  Male | 9 | 14 | 23
Region of Enrollment [Number; unit: participants]
  Japan | 21 | 43 | 64

OUTCOME MEASURES:

1. Primary Outcome: Maintenance Dose of the SPM962
Description: The maintenance dose of the SPM 962 was examined based on the safety and efficacy.
Time Frame: Up to 12 weeks after dosing
Population: Subjects in the safety analysis set who entered the maintenance period
Measure: Number; unit: participants
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 17 | 40
participants
  4.5 mg | 0 | 0
  9.0 mg | 0 | 1
  13.5 mg | 0 | 5
  18.0 mg | 3 | 5
  22.5 mg | 2 | 9
  27.0 mg | 2 | 9
  31.5 mg | 2 | 3
  36.0 mg | 8 | 8

2. Secondary Outcome: Incidence and Severity of Adverse Events, Vital Signs, and Laboratory Parameters
Description: Incidence and severity of adverse events, vital signs, and laboratory parameters following the initiation of study treatment.
Time Frame: Up to 12 weeks after dosing
Population: Safety analysis set
Measure: Number; unit: participants
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 21 | 43
participants
  Any AEs | 20 | 41
  Treatment-related AEs | 19 | 36
  SAEs | 1 | 3
  Severe AEs | 1 | 1
  Discontinuation due to AEs | 5 | 5
  Death | 0 | 0
  AEs related to laboratory parameters | 7 | 8
  Discontinuation due to AEs related to labs | 0 | 1
  Clinically significant QTc prolongation | 0 | 0

3. Secondary Outcome: Total of Unified Parkinson's Disease Rating Scale (UPDRS) Part 2 Sum Score and Part 3 Sum Score for Early Parkinson's Disease Without Concomitant L-dopa Therapy
Description: Mean change (LOCF) from baseline in Total of UPDRS Part 2 sum score and Part 3 sum at 12 weeks after dosing.
  UPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 2 assesses 13 items and Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, 12 weeks after dosing
Population: Efficacy analysis set, last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 21 | 0
Scores on a scale | -8.4 (11.2) |

4. Secondary Outcome: UPDRS Part 3 Sum Score for Advanced Parkinson's Disease With Concomitant L-dopa Therapy
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 0 | 43
Scores on a scale |  | -11.7 (10.1)

5. Secondary Outcome: UPDRS Part 2 Sum Score for Early Parkinson's Disease Without Concomitant L-dopa Therapy
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 21 | 0
Scores on a scale | -1.5 (2.4) |

6. Secondary Outcome: UPDRS Part 3 Sum Score for Early Parkinson's Disease Without Concomitant L-dopa Therapy
Description: as for outcome 4
Time Frame: Baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 21 | 0
Scores on a scale | -6.9 (9.0) |

7. Secondary Outcome: UPDRS Part 2 Sum Score (on State) for Advanced Parkinson's Disease With Concomitant L-dopa Therapy.
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (on state) at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 0 | 43
Scores on a scale |  | -2.6 (3.2)

8. Secondary Outcome: UPDRS Part 2 Sum Score (Off State) for Advanced Parkinson's Disease With Concomitant L-dopa Therapy.
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (off state) at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 0 | 35
Scores on a scale |  | -4.0 (5.2)

9. Secondary Outcome: UPDRS Part 2 Sum Score (Average Score of on State and Off State) for Advanced Parkinson's Disease With Concomitant L-dopa Therapy
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (average score of on state and off state) at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 0 | 41
Scores on a scale |  | -3.2 (3.7)

10. Secondary Outcome: Total of UPDRS Part 2 Sum Score (Average Score of on State and Off State) and Part 3 Sum Score for Advanced Parkinson's Disease With Concomitant L-dopa Therapy
Description: Mean change (LOCF) from baseline in Total of UPDRS Part 2 sum score (average score of on state and off state) and Part 3 sum score at 12 weeks after dosing.
  UPDRS sub-scale Part 2 assesses 13 items and Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, 12 weeks after dosing
Population: Efficacy analysis set, LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 0 | 41
Scores on a scale |  | -14.0 (11.6)

11. Secondary Outcome: Off Time for Advanced Parkinson's Disease With Concomitant L-dopa Therapy
Description: Mean change (LOCF) from baseline in off time at 12 weeks after dosing.
Time Frame: Baseline, 12 weeks after dosing
Population: Subjects with measurable off time data at baseline and after dosing, LOCF
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Number analyzed (Participants) | 0 | 43
Hours |  | -1.98 (1.3)

ADVERSE EVENTS:
Time Frame: 5 to 13 weeks depending on maintenance dose
Arm/Group | Early-stage Parkinson's Disease | Advanced Parkinson's Disease
Serious Adverse Events (participants affected / at risk) | 1/21 | 3/43
Other Adverse Events (participants affected / at risk) | 20/21 | 41/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-stage Parkinson's Disease (N=21) | Advanced Parkinson's Disease (N=43)
Carcinoma Prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Abnormal Behaviour (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide Attempt (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early-stage Parkinson's Disease (N=21) | Advanced Parkinson's Disease (N=43)
Nausea (Gastrointestinal disorders) | 8 (9) | 9 (10)
Vomiting (Gastrointestinal disorders) | 4 (4) | 5 (8)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Administration Site Reaction (General disorders) | 16 (16) | 20 (20)
Thirst (General disorders) | 2 (2) | 2 (2)
Nasopharyngitis (Infections and infestations) | 6 (6) | 4 (4)
Blood Urea Increased (Investigations) | 3 (3) | 1 (1)
Blood Creatine Phosphokinase Increased (Investigations) | 1 (1) | 4 (4)
Blood Urine Present (Investigations) | 2 (2) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (2) | 5 (5)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5)
Somnolence (Nervous system disorders) | 4 (5) | 7 (8)
Dizziness (Nervous system disorders) | 3 (4) | 3 (3)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 5 (5)
Dizziness Postural (Nervous system disorders) | 2 (2) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 3 (3)
hypoesthesia (Nervous system disorders) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 4 (4) | 4 (4)
Hallucination Visual (Psychiatric disorders) | 0 (0) | 4 (4)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No